CLINICAL TRIAL: NCT06355869
Title: Repeatability of Gait of Children With Spastic Cerebral Palsy in Different Walking Conditions
Brief Title: Repeatability of Gait Deviations in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s65337
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Spastic Cerebral Palsy
Keywords: Cerebral Palsy; Rehabilitation; Gait analysis; Variability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ambulatory children with spastic CP: Ambulant children with cerebral palsy between 6 and 17 years old with a consistent gait pattern. They have prescribed ankle-foot orthoses by the medical team as part of the standard care.
  Interventions: Other: repeated 3D gait-analysis
- TD children: Our TD-database of the Clinical Motion Analysis Laboratory (CMAL) of UZ Leuven was used for the calculation of the gait indices.

INTERVENTIONS:
Other: repeated 3D gait-analysis — An observational 3D gait-analysis was performed with a period of 1-14 days is foreseen between the two measurements.
  Groups: Ambulatory children with spastic CP

SUMMARY:
Three-dimensional gait analysis (3DGA) is the 'gold standard' for measurement and description of gait. Gait variability can arise from intrinsic and extrinsic factors and may vary between walking conditions. This study aimed to define the inter-trial (intrinsic) and inter-session (extrinsic) repeatability in gait analysis data of children with CP who were walking in four conditions, namely barefoot or with ankle-foot orthosis, and overground or treadmill.

DETAILED DESCRIPTION:
With a prevalence of two to three per 1000 live births, Cerebral Palsy (CP) is the most common motor disability of childhood. Improving disturbed gait in ambulatory children with CP is an important treatment goal because it is associated with functional independence and participation of children in the society. It is a common practice to prescribe ankle-foot orthoses (AFO) for ambulatory children to improve their gait, prevent secondary deformities, provide an improved base of support, and compensate for muscle weakness.

Three-dimensional gait analysis (3DGA) is the 'gold standard' for measurement and description of gait. However, gait variability can arise from intrinsic (i.e., caused by the person's natural gait variability) and extrinsic (i.e., methodological sources, such as marker placement errors) factors and may vary between walking conditions. Follow-up and/or pre- and post-intervention 3DGA's are used to determine the treatment for these children with CP. So, it is important to know when differences between 3DGA's can be seen as 'true differences' or when the difference can be explained by intrinsic/extrinsic gait variability.

The purpose of the current study is to quantify the repeatability of gait in children with CP. Therefore, the repeatability between two 3DGA's that are performed at the Clinical Motion Analysis Laboratory (CMAL) of UZ Leuven will be assessed, following the standard 3DGA procedure that is applied at CMAL for routine clinical follow-up.

On the first test day, subjects will first receive a standard clinical examination preceding the clinical overground 3DGA that is planned as a routine clinical follow-up at the CMAL, extended with an additional 3DGA on the treadmill. The treadmill gait laboratory and overground gait laboratory are across the hall from each other, which makes it possible for the subject to walk from one to the other gait laboratory in just a minute.

On the second test day, a repeated 3DGA overground and on the treadmill will be performed by the same clinician. This involved clinical assessor is well-trained to perform 3GDA in children with CP.

Between the measurements, a period from 1 - 14 days is foreseen. The combinations of repeated gait trials per test day, and the repeated test days, with involvement of only one assessor, facilitates the distinction between intrinsic and extrinsic variability.

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Function Classification System (GMFCS) level I - III
* CP (bilateral & unilateral)
* Age: 6 - 17 years
* Prescribed AFO by the medical team (as part of the standard care)

Exclusion Criteria:

* Severe contractures or spasticity, which makes it impossible to wear a conventional AFO
* Cognitive or visual impairment that hinder them to understand instructions
* Previous surgery on bones and/or muscles of the legs in the last 12 months prior to assessment
* Presence of ataxia or dystonia

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ambulant children with cerebral palsy between 6 and 17 years old with a consistent gait pattern. They have prescribed ankle-foot orthoses by the medical team as part of the standard care.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The standard error of measurement (SEM) of the continuous kinematic gait waveforms | A period of 1-14 days is foreseen between the two measurements (3DGA)
  The SEM, is the standard deviation of a number of measurements made on the same participant.
  SEM= √((∑▒〖deviations^2 〗)/(degrees of freedom)). The primary advantage of the SEM lies in providing a direct indication of measurement error in the same units as the original measurement. This characteristic makes the use of SEM particularly clinically relevant. The SEM was used as a statistical analysis for determining the inter-trial and -session variability of the kinematic continuous waveforms in the sagittal plane of the hip, knee and ankle joint. Thereby, the SEM was calculated timepoint-by-timepoint from the continues waveforms, according to the methods of Schwartz et al. [4]
The intra-class correlation (ICC) of the gait indices | A period of 1-14 days is foreseen between the two measurements (3DGA)
  The inter-trial and -session variability was defined by the use of the intra-class correlation coefficient (ICC; 2,1) (two-way random model with absolute agreement), along with the 95% confidence interval of the gait indices (i.e., the gait profile score and the gait variable score of the hip flexion, the knee flexion and the ankle dorsiflexion).
The standard error of measurement (SEM) of the continuous kinetic gait waveforms | A period of 1-14 days is foreseen between the two measurements (3DGA)
  The SEM, is the standard deviation of a number of measurements made on the same participant.
  SEM= √((∑▒〖deviations^2 〗)/(degrees of freedom)). The primary advantage of the SEM lies in providing a direct indication of measurement error in the same units as the original measurement. This characteristic makes the use of SEM particularly clinically relevant. The SEM was used as a statistical analysis for determining the inter-trial and -session variability of the kinetic continuous waveforms (i.e., moments & powers) in the sagittal plane of the hip, knee and ankle joint. Thereby, the SEM was calculated timepoint-by-timepoint from the continues waveforms, according to the methods of Schwartz et al. [4]
The standard error of measurement (SEM) of the gait indices | A period of 1-14 days is foreseen between the two measurements (3DGA)
  The SEM, is the standard deviation of a number of measurements made on the same participant. SEM= SD x √(1-ICC), where SD is the standard deviation of the grand mean (mean of session 1 and session 2) from all participants. The SEM was calculated for the gait indices (i.e., the gait profile score and the gait variable score of the hip flexion, the knee flexion and the ankle dorsiflexion).
  The primary advantage of the SEM lies in providing a direct indication of measurement error in the same units as the original measurement, which makes the use of SEM particularly clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, prof. dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Background] Sankar C, Mundkur N. Cerebral palsy-definition, classification, etiology and early diagnosis. Indian J Pediatr. 2005 Oct;72(10):865-8. doi: 10.1007/BF02731117. PMID 16272660
- [Background] Morris C, Bowers R, Ross K, Stevens P, Phillips D. Orthotic management of cerebral palsy: recommendations from a consensus conference. NeuroRehabilitation. 2011;28(1):37-46. doi: 10.3233/NRE-2011-0630. PMID 21335676
- [Background] Schwartz MH, Trost JP, Wervey RA. Measurement and management of errors in quantitative gait data. Gait Posture. 2004 Oct;20(2):196-203. doi: 10.1016/j.gaitpost.2003.09.011. PMID 15336291
- [Derived] Everaert L, Dewit T, Huenaerts C, Van Campenhout A, Labey L, Desloovere K. Repeatability of gait of children with spastic cerebral palsy in different walking conditions. J Biomech. 2024 Nov;176:112301. doi: 10.1016/j.jbiomech.2024.112301. Epub 2024 Aug 31. PMID 39265255